CLINICAL TRIAL: NCT06201728
Title: The Role of Asthma Flare-up Clinic in Improving Management and Outcomes of Asthma
Brief Title: The Effect of Asthma Flare-up Clinic After Exacerbation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0714-23-TLV
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Asthma; Asthma Attack
Keywords: Asthma flare-up; Asthma management; clinic; pulmonologist
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: For inclusion, each week, all patients that were discharged from the hospital an adhere to the inclusion criteria will be identified using an electronic medical records software (Chameleon) and a list with their details will be created. The diagnosis of asthma and of the exacerbation will be verified by senior pulmonologist. Following that, the research coordinator will contact each subject with details on the study and a preliminary acceptance for inclusion. After acceptance, the randomization will be performed manually by randomly choosing from 200 identical envelops (100 with printed "intervention" and 100 with "control").
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will include 3 follow-up visits in the flare up clinic - one month after hospital discharge (from ED or admission), 3 months after the first visit, 6 months after the second visit. At 12 and 18 months after the first visit there will be an additional phone-call with structured interview.
  Each clinic visit will include:
  i. Pulmonologist examination, review of disease state and care, and adjustment of treatment.
  ii. Vital signs (blood pressure, saturation in room air, pulse). iii. Blood sample for complete blood count. iv. Filling Asthma Quality of Life Questionnaire (AQLQ). v. Spirometry. vi. Impulse oscillometry and FeNO tests. vii. Arrangement of next follow-up visit.
  Interventions: Other: Follow-up in a flare-up clinic
- Control (No Intervention): The control group will undergo 4 phone-call follow-ups with structured interview based on a predefined questionnaire, at the following time frames - 1, 4, 10, 13, and 19 months after hospital discharge.
  Each follow-up call will include:
  i. Assessment of ACT score. ii. Whether they attend pulmonologist follow-up visit, additional evaluations (IOS or spirometry), and interventions (pulmonary rehabilitation and smoking cessation programs).
  iii. Current treatment. iv. Asthma exacerbations, use of systemic steroids, and relevant management.

INTERVENTIONS:
Other: Follow-up in a flare-up clinic — Follow-up in the clinic based on the time frame specified above. Additional interventions during the clinic visit, other than specified above, includes: An overview by a pulmonologist of new exacerbations, systemic steroid use, or other hospitalizations, active medications and compliance to treatment, inhaler using technique, possible medication side-effects, and the asthma control test (ACT) score. The physician will provide information on smoking cessation when relevant and pulmonary rehabilitation. In addition, decision on change of treatment and further evaluations outside of the clinic, including initiation of biologic treatment.
  Arms: Intervention

SUMMARY:
The goal of this interventional study is to examine the effect of asthma flare-up clinic follow-up in adult subjects after an asthma flare-up. This study aim to answer the following questions:

1. Does a follow-up in a flare-up clinic improves disease outcomes?
2. Does a follow-up in a flare-up clinic improves disease management?

Participants in the intervention group will take part in a structured follow-up at the asthma flare-up clinic at three time points. Each visit will include questionnaires, pulmonologist examination and consultation, laboratory tests and spirometry. The control group will undergo phone-call follow-up with a research coordinator in similar time frames as the intervention.

Researchers will compare the two groups to see if the clinic follow-up affects the study outcomes.

DETAILED DESCRIPTION:
The primary outcomes will be analyzed as total exacerbations during the time frame and as a time-dependent variable (time to exacerbation) using Kaplan Meier survival analysis. Additional sub-analyses will be made for the type of inclusion setting (ED/hospitalization), number of prior exacerbations, and eosinophil count. Additional analyses will be made for all secondary outcomes. Analyses relevant only for the intervention group (such as spirometry and IOS) will compare results to the first follow-up visit. A cost-effectiveness analysis will be made, comparing the follow-up cost and the cost saved by exacerbation reduction based on the final results.

Sample size calculation - The invetigators assume based on previous research that the intervention will lead to a 20% decrease in exacerbations during the 12 months from first follow-up. To achieve an alpha of 0.05 and a power of 80%, there is a need for 88 patients in each group. Assuming a loss-to-follow-up rate (missing to complete at least 2 clinic visits or loss to phone follow-up) of 20%, the study will need 115 patients in each group (230 overall).

ELIGIBILITY:
Inclusion Criteria:

* Prior asthma diagnosis based on clinical and spirometry accepted criteria.
* Acute exacerbation of asthma as the main reason for ED arrival.
* Ability to perform in-person and telephone follow-up.
* Agree to participate, with a signed or verbal informed consent, according to the study group.

Exclusion Criteria:

* Uncontrolled comorbidity.
* Cognitive dysfunction.
* Patients under 18 years or above 75 years.
* Chronic obstructive pulmonary disease (COPD) or other lung diseases (eg, idiopathic pulmonary fibrosis, Churg-Strauss Syndrome, etc) which may impair lung function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Exacerbations | During study follow-up (12 months from inclusion)
  The rate of severe asthma exacerbations between the intervention and control, defined as a deterioration of asthma leading to treatment for 3 days or more with systemic glucocorticoids or hospitalization or an emergency department visit leading to treatment with systemic glucocorticoids.

SECONDARY OUTCOMES:
Hospital arrival | During study follow-up (12 months from inclusion)
  The rate of asthma exacerbations leading to hospital arrival between the intervention and control
Systemic steroids | During study follow-up (12 months from inclusion)
  The rate of systemic steroids use between the intervention and control
Asthma control score | During study follow-up (12 months from inclusion)
  Change in asthma control score between the intervention and control. Values range 5-25, with higher scores indicating better control.
Quality of life score | During study follow-up (12 months from inclusion)
  Change in Asthma Quality of Life Questionnaire score in the intervention group. Values range 7-224, with higher scores indicating better quality of life
Time to first exacerbation | During study follow-up (12 months from inclusion)
  Time to first asthma exacerbation between the intervention and control
Time to first hospital arrival | During study follow-up (12 months from inclusion)
  Time to first hospital arrival due to asthma exacerbation and from any cause between the intervention and control
Time to first systemic steroids use | During study follow-up (12 months from inclusion)
  Time to first systemic steroid use due to respiratory symptoms between the intervention and control
Clinical remission | During study follow-up (18 months from inclusion)
  Rate of clinical remission for at least 12 months, defined as a period without exacerbations, need of systemic steroids, and an ACT above or equal to 20.
Extended clinical remission | During study follow-up (18 months from inclusion)
  Rate of extended clinical remission for at least 12 months, defined as above, with additional spirometry criteria - FEV1 after bronchodilators equal/above 80% or increase of 100 ml of pre-bronchodilator FEV1 from baseline.
Percentage of Participants with errors of inhaler use technique | During study follow-up (18 months from inclusion)
  Errors of inhaler use technique in the intervention group between clinic visits
Percentage of Participants with a change in treatment | First clinic visit (1 month after inclusion)
  Change in treatment at the first clinic visit in the intervention group
Adherent to treatment guidelines | During study follow-up (18 months from inclusion)
  Treatment adhere to the Global Initiative for Asthma (GINA) guidelines based on disease severity, in the intervention vs. the control.
Percentage of Participants with treatment compliance | During study follow-up (18 months from inclusion)
  Compliance of inhaler treatment between the intervention and control
Change in spirometry variables | During study follow-up (12 months from inclusion)
  Change in spirometry variables in the intervention group, including forced expiratory volume (FEV1) in liters and %predicted, Forced vital capacity (FVC) in liters and %predicted.
Change in FeNO results | During study follow-up (12 months from inclusion)
  Change in exhaled nitric oxide test results (FeNO) in the intervention group, in parts per billion.
Change in area of reactance using IOS | During study follow-up (12 months from inclusion)
  Change in the area of reactance (AX) using Impulse oscillometry.
Change in resonant frequency using IOS | During study follow-up (18 months from inclusion)
  Change in the reactance resonant frequency (RF, measured in Hz) using Impulse oscillometry.
Changes in respiratory resistance at 5 Hz, 20 Hz and the difference between 5 and 20 Hz using IOS | During study follow-up (12 months from inclusion)
  Change in respiratory resistance at 5 Hz (R5, measured in kPa/L/s) and 20 Hz (R20, measured in kPa/L/s), the difference between R5 and R20 (R5-R20, measured in kPa/L/s) using Impulse oscillometry.
Changes in reactance at 5 Hz using IOS | During study follow-up (12 months from inclusion)
  Change in the reactance at 5 Hz (X5) using Impulse oscillometry.

OTHER OUTCOMES:
asthma control test score - intervention | at inclusion and end of study among the intervention group.
  Asthma control test score. Values range 5-25, with higher scores indicating better control.
Analysis according to absolute peripheral eosinophils count | During study follow-up (18 months from inclusion)
  Analysis of the primary outcome base on eosinophil levels above or below 300 and 150 (as measured prior to study inclusion without steroid treatment).
Exacerbations - pre-post | comparison during the intervention to the similar time frame before inclusion
  The rate of severe asthma exacerbations, defined as a deterioration of asthma leading to treatment for 3 days or more with systemic glucocorticoids or hospitalization or an emergency department visit leading to treatment with systemic glucocorticoids.
Systemic steroids - pre-post | comparison during the intervention to the similar time frame before inclusion
  The rate of systemic steroids use
Hospital admission - pre-post | comparison during the intervention to the similar time frame before inclusion
  The rate of asthma exacerbations leading to hospital arrival between the intervention and control
Post-HOC analysis - exacerbations | At the extended duration from clinic follow-up - at 18 months
  Asthma exacerbations between the intervention and control groups
Post-HOC analysis - hospital arrival due to asthma exacerbation | At the extended duration from clinic follow-up - at 18 months
  Rate of hospital arrival due to asthma exacerbation between the intervention and control group
Post-HOC analysis - ACT score | At the extended duration from clinic follow-up - at 18 months
  Changes in the Asthma control test score (ACT) between the intervention and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDonald VM, Gibson PG. Exacerbations of severe asthma. Clin Exp Allergy. 2012 May;42(5):670-7. doi: 10.1111/j.1365-2222.2012.03981.x. PMID 22515389
- [Background] Mincheva R, Ekerljung L, Bossios A, Lundback B, Lotvall J. High prevalence of severe asthma in a large random population study. J Allergy Clin Immunol. 2018 Jun;141(6):2256-2264.e2. doi: 10.1016/j.jaci.2017.07.047. Epub 2017 Sep 20. PMID 28939411
- [Background] Naqvi M, Khachi H. The barriers to accessing primary care resulting in hospital presentation for exacerbation of asthma or chronic obstructive pulmonary disease in a large teaching hospital in London. Respir Med. 2016 Aug;117:162-5. doi: 10.1016/j.rmed.2016.05.020. Epub 2016 May 27. PMID 27492527
- [Background] Zhang X, Lai Z, Qiu R, Guo E, Li J, Zhang Q, Li N. Positive change in asthma control using therapeutic patient education in severe uncontrolled asthma: a one-year prospective study. Asthma Res Pract. 2021 Jul 21;7(1):10. doi: 10.1186/s40733-021-00076-y. PMID 34289896
- [Background] Hsu J, Wilhelm N, Lewis L, Herman E. Economic Evidence for US Asthma Self-Management Education and Home-Based Interventions. J Allergy Clin Immunol Pract. 2016 Nov-Dec;4(6):1123-1134.e27. doi: 10.1016/j.jaip.2016.05.012. Epub 2016 Sep 19. PMID 27658535
- [Background] Goeman D, Jenkins C, Crane M, Paul E, Douglass J. Educational intervention for older people with asthma: a randomised controlled trial. Patient Educ Couns. 2013 Dec;93(3):586-95. doi: 10.1016/j.pec.2013.08.014. Epub 2013 Aug 19. PMID 24007766